CLINICAL TRIAL: NCT00172263
Title: The Interaction Between Severe Acute Respiratory Distress Syndrome Viral Proteins and Monocytes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 9261701054
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Severe Acute Respiratory Syndrome
Keywords: Immunology
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: blood sampling

SUMMARY:
Severe acute respiratory syndrome (SARS) is a new threat to public health since November, 2002. The SARS is highly contagious and is believed to be transmitted by person-to-person through droplet and direct contact. The patients present with fever, chills, cough, myalgia, dyspnea, and diarrhea. The symptoms aggravate in the second week and nearly 40% of the patients develop respiratory failure that requires assisted ventilation. The mortality rate is reported as 6.5%-7%.

After several months, the world scientists found the etiology to be a new coronavirus not belonging to the previous coronavirus group I, II and III. The new virus is called SARS associated coronavirus (SARS-CoV).

Although the high morbidity and mortality of SARS occurred in adults, there was rare mortality reported in the children. The report from Hong Kong pointed out that the symptoms of SARS in younger children were milder and the clinical course was not as aggressive as in adults. Therefore, the aim of the project is to design the experiment to see the differences of immunological responses to SARS-CoV protein in healthy younger children, teenagers, and adults. The investigators hope that the result could explain the reason for milder disease in younger children and the immunological pathogenesis of SARS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, children and cord blood

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chieh Wang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Li-Chieh Wang, MD, Taipei, Taiwan, China